CLINICAL TRIAL: NCT03822260
Title: Comparasion of Bio-markers and Neuroimaging Changes Caused by Neuroenflamation After the Aneurysmal Subarachnoid Hemorrhage
Brief Title: Evaluation of Neuroinflamation of SAH
Acronym: BAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: TD -001
Record Dates: First submitted 2018-11-12; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — In the blood plasma stored in the temperature of -86 'C for the period not longer than 6 months, the concentration of the following parameters was marked with the use of immunoenzymatic ELISA method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sur1/ Trpm 4 acitivities at SAH: only after collecting sample,
  Interventions: Diagnostic Test: Bezmialem VAkif Unv. Ethical board

INTERVENTIONS:
Diagnostic Test: Bezmialem VAkif Unv. Ethical board — If ıs any trials not convenient to Helsinki Agrement about Human research rules

SUMMARY:
The investigators are planning that can these markers be used a predictive marker at SAH and for this aim we will study both patiens' blood sample and their CT image.

DETAILED DESCRIPTION:
An ideal marker which could be used clinically should meet numerous criteria, such as high sensitivity or the possibility of easy and quick assessment of its concentration in blood or blood plasma.The Fisher's scale presents an alternative for evaluating patients with subarachnoid hemorrhage . The investigator are going to evaluate both plasma markers and fishers scale at SAH.

ELIGIBILITY:
Inclusion Criteria:

* Ruptured Subarachnoid Aneursym

Exclusion Criteria:

* without aneursymal sah
* Patient's positive for rheumatoid factor and anti-CCP or with chronic inflammatory diseases (such as ankylosing spondylitis or rheumatoid arthritis), systemic diseases (such as hypercholesterolemia, hypertension, diabetes mellitus, myocardial infarction, stroke, peripheral artery disease), active infection, a history of term medication, trauma to the hip and smoking were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the emergency room of the universty hospital with aSAH have a CBC and blood sample performed on admission. Blood samples are obtained significant days (1,4-14 days) thereafter during their hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic marker identification | 24 months
  Evaluation of the concentration levels of enflamation markers relation with Sur1 TRPM+ molecules, together with the values of global tests of coagulation system, may serve as a helpful SAH diagnostic marker.

IPD SHARING:
Plan to Share IPD: Undecided
ıt was not decided